CLINICAL TRIAL: NCT01563965
Title: Effects of the Abbreviation of Preoperative Fasting With Carbohydrates and Hydrolized Proteins on the Inflammatory Response and Insulin Resistance After Major Abdominal Operations
Brief Title: Carbohydrates and Proteins 3h Before Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Jose Eduardo de Aguilar-Nascimento, MD, PhD, Federal University of Mato Grosso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pexe_aguilar; 471206/2009-1 (Other Grant/Funding Number: CNPq - Brazil 471206/2009-1)
Record Dates: First submitted 2012-03-24; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Surgery; Postoperative Complications; Inflammation
Keywords: Preoperative fasting; Acute phase proteins; Carbohydrates; Protein hydrolizate; Inflammatory response; Surgery
MeSH Terms: conditions — Postoperative Complications; Inflammation | interventions — Carbohydrates; Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional preoperative fast (Active Comparator): Patients underwent surgery after 8h fast
  Interventions: Other: Preoperative fasting of 8h
- Carbohydrate plus protein beverage (Experimental): The study group received 400 ml (evening drink) or 200 ml (3h prior to operation drink) of a solution containing 11% de protein (pea hydrolized proptein), 89% de carbohydrates (maltodextrin 79% and saccharose 21%) e 0% of lipids (Providextra, Fresenius Kabi, São Paulo, Brasil).All the patients fasted for solids at least 8 hours from the operation
  Interventions: Dietary Supplement: Carbohydrate plus hydrolyzed protein beverage

INTERVENTIONS:
Dietary Supplement: Carbohydrate plus hydrolyzed protein beverage — The study group received 400 ml (evening drink) or 200 ml (3h prior to operation drink) of a solution containing 11% de protein (pea hydrolized proptein), 89% de carbohydrates (maltodextrin 79% and saccharose 21%) e 0% of lipids (Providextra, Fresenius Kabi, São Paulo, Brasil). All the patients fasted for solids at least 6 hours from the operation
  Other Names: Providextra, Fresenius Kabi, São Paulo, Brasil
  Arms: Carbohydrate plus protein beverage
Other: Preoperative fasting of 8h — Conventional protocol of 8h fasting before an operation
  Other Names: Control group
  Arms: Conventional preoperative fast

SUMMARY:
Prolonged pre-operative fasting increases postoperative hospital stay and current evidence recommends carbohydrate (CHO) drinks 2 hours before surgery. Our hypothesis is that the addition of hydrolized protein to a CHO-based drink not only reduces the inflammatory response but also diminish hospitalization.

DETAILED DESCRIPTION:
This was a randomized, double-blind, clinical study carried out at the Julio Muller University Hospital (Mato Grosso State, Brazil). The study was approved by the hospital Research Ethics Committee registered under number 723/CEP-HUJM/09 and is in accordance with the ethics principals set out in the Helsinki Declaration (2000), and meets Brazilian national legal specifications.

Inclusion criteria includes adults (18-65 years-old), of both sexes, and candidates to elective major operations such as subtotal gastrectomy, colectomy, and anterior resection of the rectum for malignancies. Exclusion criteria were having diabetes mellitus, chronic kidney failure, chronic liver disease or serum bilirubin greater than 2 mg/dL, body mass index (BMI) above 35Kg/m2, American Anesthesiologists Association (ASA) score above 3, gastro-esophageal reflux, gastroparesis or intestinal obstruction. Patients with any non-compliance with the study protocol, or who had associated operations, or presented severe intraoperative complications (any type of shock, cardiac arrest, coagulations problems), or experienced prolonged operations (lasting more than 6 hours) were also excluded.

Patient randomization was carried out on admission to the hospital using random numbers issued by a computer program (www.graphpad.com). For the randomization the precepts of the CONSORT flow diagram were followed.

The patients were randomized into two groups: the study group and the control group. The patients were given a specific drink to their group on the evening prior to surgery and three hours before the operation. The study group received 400 ml (evening drink) or 200 ml (3h prior to operation drink) of a solution containing 11% de protein (pea hydrolized proptein), 89% de carbohydrates (maltodextrin 79% and saccharose 21%) e 0% of lipids (Providextra, Fresenius Kabi, São Paulo, Brasil) and the control group received conventional 6-8h fast. All the patients fasted for solids at least 6 hours from the operation.

On the day before the surgery and on the second postoperative day blood samples were collected for glucose, insulin, triglycerides, albumin, pre-albumin, CRP, and α-1-acid glycoprotein (α-1-GA) assays. The HOMA-IR (Homeostasis Model Assessment-Insulin Resistance) equation was used to assess insulin resistance according to the formula: HOMA-IR = insulin (µU/mL) x glycaemia (mg/dL) / 405. To assess inflammatory activity the PINI (CRP (mg/L) x α-1-GA (mg/L)/ albumin (g/L) x pre-albumin (mg/L) and the CRP/albumin ratio were used.

The mean outcome variable was the length of postoperative stay. Other endpoints included the infectious morbidity, the insulin resistance assessed by HOMA-IR, and the inflammatory indexes or markers mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-65 years-old),
* of both sexes, and candidates to elective major operations such as subtotal gastrectomy, colectomy, and anterior resection of the rectum for malignancies

Exclusion Criteria:

* Diabetes mellitus,
* chronic kidney failure,
* chronic liver disease or serum bilirubin greater than 2 mg/dL,
* body mass index (BMI) above 35Kg/m2, American Anesthesiologists Association (ASA) score above 3,
* gastro-esophageal reflux,
* gastroparesis or intestinal obstruction.
* Patients with any non-compliance with the study protocol, or who had associated operations, or presented severe intraoperative complications (any type of shock, cardiac arrest, coagulations problems), or experienced prolonged

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Length of postoperative hospital stay | 12 months
  We compared the length of hospital postoperative stay in the 2 groups of the study.

SECONDARY OUTCOMES:
Inflammatory markers | 12 months
  On the day before the surgery and on the second postoperative day blood samples were collected for albumin, pre-albumin, CRP, and α-1-acid glycoprotein (α-1-GA) assays. To assess inflammatory activity the prognostic inflammatory and nutritional index (PINI)(CRP (mg/L) x α-1-GA (mg/L)/ albumin (g/L) x pre-albumin (mg/L) and the CRP/albumin ratio were calculated and used to compare the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Jose E Aguilar-Nascimento, MD, PhD, Principal Investigator — University of Mato Grosso
Locations (1):
- Hospital Universitario Julio Mullar, Cuiabá, Mato Grosso, Brazil

REFERENCES:
- [Background] Dock-Nascimento DB, de Aguilar-Nascimento JE, Magalhaes Faria MS, Caporossi C, Slhessarenko N, Waitzberg DL. Evaluation of the effects of a preoperative 2-hour fast with maltodextrine and glutamine on insulin resistance, acute-phase response, nitrogen balance, and serum glutathione after laparoscopic cholecystectomy: a controlled randomized trial. JPEN J Parenter Enteral Nutr. 2012 Jan;36(1):43-52. doi: 10.1177/0148607111422719. PMID 22235107
- [Background] Perrone F, da-Silva-Filho AC, Adorno IF, Anabuki NT, Leal FS, Colombo T, da Silva BD, Dock-Nascimento DB, Damiao A, de Aguilar-Nascimento JE. Effects of preoperative feeding with a whey protein plus carbohydrate drink on the acute phase response and insulin resistance. A randomized trial. Nutr J. 2011 Jun 13;10:66. doi: 10.1186/1475-2891-10-66. PMID 21668975
- [Background] de Aguilar-Nascimento JE, Dock-Nascimento DB. Reducing preoperative fasting time: A trend based on evidence. World J Gastrointest Surg. 2010 Mar 27;2(3):57-60. doi: 10.4240/wjgs.v2.i3.57. PMID 21160851